CLINICAL TRIAL: NCT03790839
Title: A Phase 1, Open-Label, Sequential, Multiple-Dose, Drug-Drug Interaction Study of Dorzagliatin and Sitagliptin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Drug Interaction Study Between Dorzagliatin and Sitagliptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMM0111
Record Dates: First submitted 2018-12-27; First posted 2019-01-02 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2018-12

CONDITIONS: Patients
MeSH Terms: interventions — Sitagliptin Phosphate; Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential arm ABC (Experimental): A: Sitagliptin 100 mg QD in the morning on Days 1-5; B: Sitagliptin 100 mg QD in the morning and dorzagliatin 75 mg BID (morning and evening) on Days 6-10, with only the morning dose on Day 10; C: Dorzagliatin 75 mg BID (morning and evening) on Days 11-15, with only the morning dose on Day 15.
  Interventions: Drug: Sitagliptin; Drug: Dorzagliatin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin (Januvia® 100 mg tablets for oral administration)
  Other Names: Januvia
Drug: Dorzagliatin — Glucokinase activator currently under development
  Other Names: HMS5552

SUMMARY:
This is a Phase 1, open-label, sequential, multiple-dose, drug interaction study of glucokinase activator dorzagliatin and sitagliptin in subjects with T2DM. Pharmacokinetics and pharmacodynamics when dorzagliatin and sitagliptin given alone and in combination will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with T2DM within at least 3 months prior to screening
2. Male and/or female subjects between the ages of 30 and 65 years, inclusive;
3. Body Mass Index (BMI) of 19 to 38 kg/m2, inclusive;
4. Fasting C-peptide test result >0.3 nmol/L (>0.90 ng/mL);
5. HbA1c ≥7% and ≤10.5%;

Exclusion Criteria:

1. Fasting blood glucose at screening or Day -1 ≤110 or ≥270 mg/dL;
2. Type 1 diabetes mellitus;
3. Reported incidence of severe or serious hypoglycemia within 3 months prior to screening;
4. Known contraindications to sitagliptin;
5. Clinically significant gastrointestinal disorder;
6. History or symptoms of clinically significant cardiovascular disease within one year prior to screening;
7. History of more than three urinary tract infections and/or more than three genital fungal infections in the last 12 months;
8. Reported history of clinically significant central nervous system disease;
9. Reported history of liver disease;
10. Reported history of clinically significant renal disease;
11. Estimated glomerular filtration rate (eGFR) ≤60 mL/min/1.73m2;
12. Acute or chronic metabolic acidosis, including diabetic ketoacidosis;
13. Known or suspected malignancy;
14. Any reported hypersensitivity or intolerance to sitagliptin;
15. Antidiabetic treatment with insulin, sulfonylureas, thiazolidinediones or GLP-1 agonist within 3 months prior to screening;
16. Systolic blood pressure <90 or >160 mmHg or diastolic blood pressure <60 or >100 mmHg at screening;
17. A hospital admission or major surgery within 90 days prior to screening;
18. Uncontrolled hypertriglyceridemia >500 mg/dL;
19. Positive blood screen for HIV, hHBsAg, or hepatitis C antibody;
20. Positive pregnancy test result;
21. Female is breast-feeding or planning to become pregnant;
22. Treated with any investigational drugs within 6 weeks prior to screening;
23. Reported history of prescription drug abuse;
24. Reported history of alcohol abuse;
25. Reported history of donation or or acute loss of blood during the 90 days prior to screening;

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Geometric mean ratio (GMR) for Cmax of sitagliptin | up to 10 days
  GMR between combination and sitagliptin monotherapy for Cmax of sitagliptin
GMR for AUC0-24h of sitagliptin | up to 10 days
  GMR between combination and sitagliptin monotherapy for AUC0-24h of sitagliptin
GMR for Cmax of dorzagliatin | up to 15 days
  GMR between combination and dorzagliatin monotherapy for Cmax of dorzagliatin
GMR for AUC0-24h of dorzagliatin | up to 15 days
  GMR between combination and dorzagliatin monotherapy for AUC0-24h of dorzagliatin
Adverse events | up to 15 days
  Number of participants with AEs
Abnormal vital signs | up to 15 days
  Number of participants with abnormal vital signs (blood pressure, pulse rate, respiratory rate and oral temperature)
Abnormal clinical laboratory findings | up to 15 days
  Number of participants with abnormal clinical laboratory findings
12-lead ECG | up to 15 days
  Number of participants with abnormal ECG VR,, PR, QRS and QT

SECONDARY OUTCOMES:
iCmax of glucose | up to 15 days
  The incremental peak plasma concentration of glucose post OGTT
iAUC0-4h of glucose | up to 15 days
  The incremental area under the concentration-time curve of glucose in 4 hours post OGTT
iCmax of C-peptide | up to 15 days
  The incremental peak plasma concentration of C-peptide post OGTT
iAUC0-4h of C-peptide | up to 15 days
  The incremental area under the concentration-time curve of C-peptide in 4 hours post OGTT
iCmax of GLP-1 | up to 15 days
  The incremental peak plasma concentration of GLP-1 post OGTT
iAUC0-4h of GLP-1 | up to 15 days
  The incremental area under the concentration-time curve of GLP-1 in 4 hours post OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tracey, MD, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services Inc., Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No